CLINICAL TRIAL: NCT01258322
Title: Twelve Weeks of Pioglitazone Therapy Significantly Attenuates Dysmetabolism and Reduces Inflammation in Prevalent Peritoneal Dialysis Patients. A Randomized, Cross-over Trial.
Brief Title: Pioglitazone Attenuates Dysmetabolism in Peritoneal Dialysis (PD) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Dr. Tongying Zhu, Huashan Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Neph-1000
Record Dates: First submitted 2010-12-09; First posted 2010-12-10 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2007-03

CONDITIONS: Peritoneal Dialysis; Pioglitazone; Hypertriglyceridemia; Insulin Resistance; Inflammation
MeSH Terms: conditions — Hypertriglyceridemia; Insulin Resistance; Inflammation | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- pioglitazone (Experimental)
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — The patients were randomized divided into 2 groups; one received no pioglitazone for lowing triglyceride, one with oral pioglitazone (Actos®, Takeda®) 15mg once daily for 12 weeks. After a four-week wash out, patients then continued with the alternate therapy.
  Other Names: pioglitazone (Actos®, Takeda®) 15mg

SUMMARY:
1. Background:Cardiovascular disease (CVD) is the major cause of mortality in peritoneal dialysis (PD) patients, in whom it is partly attributable to a higher prevalence of dysmetabolism. Currently, few treatments are available with a proven effect on dyslipidemia, insulin resistance and inflammation in this patient group.
2. Study design: Randomized, cross-over trial.
3. Settings and Participants: Prevalent PD patients (>20 years old, s-triglycerides >1.8 mmol/L) who had never received glitazones were enrolled.
4. Interventions: Participants were randomized to receive either oral pioglitazone (PIO; 15 mg once daily) and no pioglitazone, both for 12 weeks and in random order, with a four-week wash out in between.
5. Outcomes and measurements: The primary endpoint was change of serum triglyceride (TG) level during the PIO as compared to no PIO. Secondary endpoints included changes in other lipid levels, HOMA-IR, adipocytokines and CRP. Outcome effects were assessed using a GLM.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the major cause of mortality in chronic kidney disease, including peritoneal dialysis (PD) patients. While survival has not been shown to differ between peritoneal and hemodialysis, because of glucose uptake from the dialysate PD patients are more prone to dyslipidemia, insulin resistance (IR) and obesity. These metabolic disorders are substantially linked to the development of CVD and mortality in this patient population.

Hypertriglyceridemia, reported to be present in 70% of PD patients, is linked to both glucose uptake from the peritoneum and IRand promote vascular damage. Inflammation has been proposed to be a fundamental promoter of atherosclerosis and demonstrated a dose-response relationship between C-reactive protein (CRP) and mortality . Adipocytokines, such as adiponectin，leptin and resistin, also play important roles in the development of dyslipidemia, IR, atherosclerosis, inflammation and CVD in PD patients. Therefore, therapies targeted at metabolic disorder are an important component of treatment for PD patients. Fibrates, peroxisome proliferator-activated receptors (PPAR)-α agonist, can lower serum TG, however, its use in PD patients is limited by its limited efficacy and often-appeared adverse effects such as rhabdomyolysis and hepatic impairment. Nowadays, PPAR-γ agonist, thiazolidinediones (TZDs), represented by pioglitazone and rosiglitazone, exert their hypoglycemic properties through reduction of insulin resistance. For more than ten years, they have been used to control blood glucose in type 2 diabetes mellitus (T2DM). In addition, TZDs have also been noted to have beneficial effects on lipid metabolism and inflammation apart from their effects on glycogenic control. However, the study about TZDs in the treatment of metabolic disorder in PD patients, especially in nondiabetic subjects is very scarce and limited.

We, therefore set out to investigate the effect of TZDs, pioglitazone on hyperlipidemia, insulin resistance, inflammation and adipokine dysmetabolism of PD patients, especially in nondiabetic patients.

ELIGIBILITY:
Inclusion Criteria:

All patients received more than one month regular continuous ambulatory peritoneal dialysis(CAPD) or intermittent peritoneal dialysis(IPD). The causes of chronic renal failure were diabetes and non-diabetes.-

Exclusion Criteria:

history of allergy to thiazolidinediones and fenofibrate; history of any sever adverse event for fibrate that can't be tolerated by the patients; patient can not be follow-up regularly; history of myocardial infarction(MI) or coronary artery bypass graft (CABG) surgery within the past 1 month, history of cerebral vascular accident (CVA) or percutaneous transluminal coronary angioplasty(PTCA) within the past 6 months; chronic use of non-steroidal anti-inflammatory drugs(NSAIDs), steroids or immunosuppressives; patient with the acute infection; patient with malignant tumor; have the evidence of severe hepatic injury (ALT/AST>100u/L).-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
change of serum TG level | 12 weeks

SECONDARY OUTCOMES:
the change of serum CHO, LDL. HDL level, HOMA-IR, adipocytokines level and CRP | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tongying Zhu, MD and PhD, Principal Investigator — Huashan Hospital